CLINICAL TRIAL: NCT01175031
Title: Validation of Breathing Event Detection of the Philips Respironics Sleep Therapy System REMstar Auto A-Flex Compared to Clinical Polysomnography
Brief Title: Comparison of Breathing Event Detection by a Continuous Positive Airway Pressure Device to Clinical Polysomnography
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philips Respironics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ST-1002-PRS1ED-MS
Record Dates: First submitted 2010-07-30; First posted 2010-08-04 (Estimated); Results first posted 2016-05-02 (Estimated); Last update posted 2018-10-31 (Actual); Status verified 2018-10

CONDITIONS: Sleep Apnea Central; Cheyne-Stokes Respiration; Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Central; Cheyne-Stokes Respiration; Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- REMstar Auto with A-Flex (Experimental): Manipulation of positive airway pressure (PAP) will occur throughout the night to induce breaking events. PAP will be set to the participant's prescribed pressure, increased until breathing events are induced, and then returned to the prescribed pressure. This cyclic pattern will continue throughout the night. Events will be measured with REMstar Auto with A-Flex.
  Interventions: Other: Manipulation of Positive Airway Pressure (PAP)
- Manually Scored Polysomnography (PSG) (Other): Manipulation of positive airway pressure (PAP) will occur throughout the night to induce breaking events. PAP will be set to the participant's prescribed pressure, increased until breathing events are induced, and then returned to the prescribed pressure. This cyclic pattern will continue throughout the night. Events will be Manually Scored Polysomnography (PSG).
  Interventions: Other: Manipulation of Positive Airway Pressure (PAP)

INTERVENTIONS:
Other: Manipulation of Positive Airway Pressure (PAP) — Positive airway pressure (PAP) will be manipulated throughout the night to induce breathing events. PAP will be set to the participant's prescribed pressure, increased until breathing events are induced , and then returned to the prescribed pressure. This cyclic pattern will continue throughout the night.

SUMMARY:
The purpose of this study is to demonstrate diagnostic agreement and determine the accuracy of the continuous positive airway pressure (CPAP) device compared to simultaneous, attended clinical polysomnography (PSG) in identifying breathing events in participants previously diagnosed with complex sleep apnea (CompSAS), complex sleep apnea with Cheyne-Stokes respiration (CSR), or obstructive sleep apnea (OSA).

DETAILED DESCRIPTION:
Study Objectives: To compare a positive airway pressure (PAP) device's detection of respiratory events and airway status during device detected apneas with events scored on simultaneous polysomnography (PSG).

Design: Prospective PSGs of patients with sleep apnea using a new-generation PAP device.

Settings: Four clinical and academic sleep centers.

Patients: Forty-five patients with obstructive sleep apnea (OSA) and complex sleep apnea (Comp SA) performed a PSG on PAP levels adjusted to induce respiratory events.

Interventions: None.

ELIGIBILITY:
Inclusion Criteria:

* Males and females, ages 21-80.
* Able and willing to provide written informed consent.
* Diagnosis of complex sleep apnea (CompSAS) or Obstructive Sleep Apnea (OSA) within one year of study participation.
* For participants with CompSAS: (a) Diagnostic PSG with an Apnea-Hyopnea Index (AHI) greater than or equal to 10 events/hour and central apnea index (CAI) greater than or equal to 5 events/hour of sleep or (b) PAP titration with a CAI greater than or equal to 5 events/hour of sleep.
* For participants with OSA, a diagnostic PSG with an AHI greater than or equal to 15 events/hour of sleep.
* Must have had a CPAP titration such that the necessary PAP level to treat the sleep disordered breathing is known.
* Agreement to undergo a full-night, in-laboratory PSG on CPAP device.

Exclusion Criteria:

* Participation in an interventional research study within 30 days of study participation.
* Pre-menopausal females known to be pregnant or who are sexually active and not using a reliable method of birth control.
* Surgery of the upper airway, nose, sinus, or middle ear within the last 90 days.
* Surgery at any time for the treatment of OSA such as uvulopalatopharyngoplasty (UPPP).
* Major medical or psychiatric condition that would interfere with the demands of the study, adherence to positive airway pressure, or the ability to complete the study.
* Chronic respiratory failure or insufficiency with suspected or known neuromuscular disease, moderate or severe Chronic Obstructive Pulmonary Disease (COPD) or other pulmonary disorders, or any condition with an elevation of arterial carbon dioxide levels (> 45 mmHg) while awake.
* Currently prescribed oxygen therapy.
* Ventilatory induced barotrauma within 6 months of study participation.
* Untreated insomnia.
* Other major medical condition that, in the judgment of the investigator, precludes participation in this study.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2010-09; Primary Completion 2013-06 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Berry, MD, Principal Investigator — University of Florida; Sheila Tsai, MD, Principal Investigator — National Jewish Health
Locations (3):
- United States (3):
  - National Jewish Health, Denver, Colorado
  - University of Florida - Shands Sleep Disorders Center, Gainesville, Florida
  - Sleep Health, Portage, Michigan

RESULTS

PARTICIPANT FLOW:
Groups:
- Sleep Apnea: Individuals with Obstructive Sleep Apnea (OSA); Complex Sleep Apnea (CompSAS) and central apnea index (CAI), or the PSG during PAP treatment had a central apnea index ≥ 5 events/h after obstructive apneas resolved.
Period: Overall Study
Arm/Group | Sleep Apnea
Started | 45
Completed | 45
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Sleep Apnea
Number analyzed (Participants) | 45
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.2 (13.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 29
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 32
  African American | 8
  Hispanic/Latino | 2
  Others | 3
Region of Enrollment [Number; unit: participants]
  United States | 45
Body mass index [Mean (Standard Deviation); unit: kg/m^2] | 53.2 (13.9)
Diagnostic Apnea-Hypopnea Index (AHI) [Mean (Standard Deviation); unit: events/hour] | 39.3 (26.0)
Diagnosis [Number; unit: participants]
  Obstructive Sleep apnea | 32
  Complex Sleep Apnea | 13

OUTCOME MEASURES:

1. Primary Outcome: Number of Breathing Events Identified by the Continuous Positive Airway Pressure (CPAP) Device Compared to a Simultaneous Polysomnography
Description: The following breathing events: RERAs, central apneas, periodic breathing, obstructive apneas, and hypopneas in patients previously diagnosed with CompSAS or OSA detected by simultaneous Polysomnography and REMstar Auto with A-Flex were compared.
Time Frame: During a single night of polysomnography lasting an average of 8 hours
Measure: Mean (Standard Deviation); unit: events/hour
Groups:
- REMstar Auto With A-Flex; Manually Scored Polysomnography (PSG): Manipulation of positive airway pressure (PAP) will occur throughout the night to induce breaking events. PAP will be set to the participant's prescribed pressure, increased until breathing events are induced, and then returned to the prescribed pressure. This cyclic pattern will continue throughout the night. Events will be measured with REMstar Auto with A-Flex and Manually Scored Polysomnography (PSG).
  Manipulation of Positive Airway Pressure (PAP): Positive airway pressure (PAP) will be manipulated throughout the night to induce breathing events. PAP will be set to the participant's prescribed pressure, increased until breathing events are induced , and then returned to the prescribed pressure. This cyclic pattern will continue throughout the night. It will be measure by the REMstar Auto with A-Flex and manually scored PSG.
Arm/Group | REMstar Auto With A-Flex | Manually Scored Polysomnography (PSG)
Number analyzed (Participants) | 45 | 45
events/hour
  Apnea-hyopnea index | 16.5 (13.5) | 18.1 (18.6)
  Apnea index | 11.4 (9.9) | 11.5 (16.0)
  Hypopnea index | 5.1 (5.0) | 6.6 (7.5)
  Respiratory effort-related arousal (RERA) index | 2.8 (2.0) | 6.3 (7.4)
Statistical Analysis 1: Comparison: REMstar Auto With A-Flex vs Manually Scored Polysomnography (PSG); Test type: Superiority or Other; p = 0.003, signed-rank tests

2. Secondary Outcome: Device Detected Apneas as Detected by Philips Respironics (PR) System One
Description: All device-detected apneas were tabulated. Then they were broken down into obstructed airway apneas and clear airway apneas. The results are recorded below as apneas with obstructed airway and apneas with clear airway.
Time Frame: During a single night of polysomnography lasting an average of 8 hours
Population: 1097 Device Detected Apneas were detected.
Measure: Number; unit: events
Units Other Than Participants: Device Detected Events
Groups:
- Device-Detected Apneas: Device-detected apneas were classified as either Clear Airway or Obstructed Airway.
Arm/Group | Device-Detected Apneas
Number analyzed (Participants) | 45
Number analyzed (Device Detected Events) | 1097
events
  Apnea with obstructed Airway | 762
  Apnea with clear airway | 335

3. Secondary Outcome: Device-Detected Obstructed Airway Apnea Agreement
Description: Device-Detected Apneas were broken down and then reviewed with the manually scored apneas. Of the Obstructed Airway apneas they were broken down into a few different categories: Manually Scored Obstructive Apneas, Manually Scored Central Apneas, Manually Scored Hypopneas and Manually Scored RERAs.
Time Frame: During a single night of polysomnography lasting an average of 8 hours
Population: 762 Device Detected Apneas were detected.
Measure: Number; unit: events
Units Other Than Participants: Device Detected Obstructed Airway Apneas
Groups:
- Device-Detected Obstructive Airway Apneas: Of the device-detected obstructive airway apneas a comparison was done of manually scored verses device detected.
Arm/Group | Device-Detected Obstructive Airway Apneas
Number analyzed (Participants) | 45
Number analyzed (Device Detected Obstructed Airway Apneas) | 762
events
  Manually Scored Obstructive Apnea | 367
  Manually Scored Central Apnea | 159
  Manually Scored Hypopnea | 180
  Manually Scored RERA | 56

4. Secondary Outcome: Device-Detected Clear Airway Apnea Agreement
Description: Device Detected Clear Airways events were counted by the device. These events were then compared to manual PSG scoring. The manual PSG scoring determined that these were apnea events. However, the manual scoring allows for more channels to be reviewed and manual scoring was able to classify them into 4 different categories: Manually Scored Obstructive Apneas, Manually Scored Central Apneas, Manually scored hypopneas and manually scored RERAs.
Time Frame: During a single night of polysomnography lasting an average of 8 hours
Population: 335 Device Detected Clear Airway Apneas were detected.
Measure: Number; unit: events
Units Other Than Participants: Device Detected Clear Airway Apneas
Groups:
- Device-Detected Clear Airway Apneas: Device-detected apneas were classified as either Clear Airway or Obstructed Airway.
Arm/Group | Device-Detected Clear Airway Apneas
Number analyzed (Participants) | 45
Number analyzed (Device Detected Clear Airway Apneas) | 335
events
  Manually Scored Obstructive Apnea | 53
  Manually Scored Central Apnea | 209
  Manually Scored Hypopnea | 49
  Manually Scored RERA | 24

ADVERSE EVENTS:
Time Frame: Adverse events were collected from screening until visit 2, these two visits were up to 7 days apart.
Groups:
- Subjects With Sleep Apnea: Subjects aged 21 thru 80 with a diagnosis of CompSAS or OSA and able to undergo a full-night in the sleep laboratory.
Arm/Group | Subjects With Sleep Apnea
Serious Adverse Events (participants affected / at risk) | 0/45
Other Adverse Events (participants affected / at risk) | 0/45

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less